CLINICAL TRIAL: NCT01346345
Title: Aesthetic Evaluation of Two Piece 3mm Implants for Single Tooth Replacement of Maxillary Laterals and Mandibular Incisors
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Dr.Suzanne Caudry Implant Dentistry and Periodontics (Other)
Responsible Party: Suzanne Caudry, PhD, DDS, MSc, Dr. Suzanne Caudry Implant Dentistry and Periodontics
Other Study IDs: WIRB® Protocol #20101573
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-04

CONDITIONS: Recession
Keywords: Recession

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aesthetic evaluation of two piece 3mm implants for single tooth replacement of maxillary laterals and mandibular incisors

DETAILED DESCRIPTION:
PURPOSE OF THE STUDY:

The purpose of this research study is to examine the aesthetics (the appearance of the implanted tooth and gums) as well as the soft tissue loss over a three-year period. This study involves replacing a missing small front tooth with a dental implant, abutment, and crown. A titanium dental implant acts as the replacement for a tooth root. An abutment is made of titanium which is either gold or silver in color and cannot be seen; but may affect the way the gum looks. An abutment is the component that attaches the crown to the implant post. A crown (which acts as the tooth replacement) is made of metal and/or porcelain and attaches over the abutment.

The dental implant and the abutments used in this study have been approved by Health Canada and the U.S. Food and Drug Administration (FDA) for the use of replacing the small teeth in the front of the mouth.

The abutment is made in two colors (either gold or silver) and you cannot choose. For each subject this is decided by chance. You will have an equal chance of getting a gold or silver-colored attachment. You will know which color the abutment will be once you have consented to be in the study and registered. You will know the color of the abutment before the implant is placed. The abutment is covered by the crown.

You will be in this study for about three years. There will be approximately 60 subjects who will participate in this study in different centres, in Canada and the USA.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide written informed consent to participate in the study.
* 18 years or older

Site requirements:

Missing one or both maxillary lateral incisors (if missing both, then both sites must be used in the study) or Single missing mandibular incisor or Two missing mandibular incisors, not adjacent to one another (both sites must be used in the study) Aside from the missing teeth specified above, all other teeth in the sextant must be present.

A minimum of premolar occlusion is required. A minimum mesio-distal and buccal-lingual distance of 5mm is required

Exclusion Criteria:

* Rampant caries or unstable periodontal disease of the remaining dentition.
* Any systemic or local disease or condition that may compromise post-operative healing.
* Long-term use of systemic corticosteroids or other medications that may compromise post-operative healing.
* Present alcohol and/or drug abuse.
* Unable or unwilling to return for follow-up exams over a 3 year period.
* Pregnancy or lactation at time of enrollment.
* Smokers will be excluded from the subject pool.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects for this study will be recruited from the practices of the six study centers (Dr. Caudry + 5 centers from the North American PEERS group) within a period of eighteen months from commencement of the study. A total of sixty subjects (ten per center) of any gender and race aged 18 and older will be accepted provided they meet the inclusion and exclusion criteria (see page 6). Dental implants for permanent tooth replacement are not indicated for use in those under the age of 18. Vulnerable subjects will not be included.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-05; Primary Completion 2015-03 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Recession | every 12 months for 3 years
  The Astra Tech 3.0 mm 2 piece implant can be placed and restored in a 5 mm or greater bone space for a mandibular incisor or maxillary lateral incisor site (minimum 5 mm mesio-distal [side to side] bone width and 5mm bucco-lingual [front to back] bone width) without exhibiting recession of the soft tissue (gingival margin or the interproximal papillae).

SECONDARY OUTCOMES:
Esthetic parameter Scores | every 12 months up to three years
  Esthetic parameter scores will be higher when the Atlantis Gold Hue titanium abutment is used in comparison to the Atlantis titanium abutment.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Suzanne D Caudry, DDS PhD, Principal Investigator — Implant Dentistry and Periodontics
Locations (1):
- Dr. Suzanne Caudry PhD DDS MSc Perio Implant Dentistry and Periodontics, Toronto, Ontario, Canada